CLINICAL TRIAL: NCT05737628
Title: First-in-human Dose Escalation and Expansion Study With the SIRPα-directed Monoclonal Antibody BYON4228 Alone and in Combination With Rituximab to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics and Efficacy in Patients With Relapsed/Refractory CD20 Positive B-cell Non-Hodgkin's Lymphoma (NHL)
Brief Title: First-in-human Dose Escalation and Expansion Study With the SIRPα-directed Monoclonal Antibody BYON4228
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Byondis B.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BYON4228.001
Record Dates: First submitted 2023-02-08; First posted 2023-02-21 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Lymphoma
Keywords: mAB; Monoclonal antibody; Lymphoma; Non-Hodgkin's Lymphoma; SIRPα; NHL; CD20; CD47; SIRP; MCL; FL; MZL; DLBCL
MeSH Terms: conditions — Lymphoma; Lymphoma, Non-Hodgkin | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BYON4228 + Rituximab (Experimental)
  Interventions: Drug: BYON4228 + Rituximab

INTERVENTIONS:
Drug: BYON4228 + Rituximab — BYON4228 is a humanized monoclonal antibody (mAb) directed against SIRPα. BYON4228 IV infusion every four weeks until disease progression or unacceptable toxicity. Different doses.
  Rituximab IV infusion (375 mg/m2) starting from the second treatment cycle onwards. Weekly infusion during the first cycle and every four weeks in subsequent 5 cycles.
  Other Names: Truxima

SUMMARY:
This is the first-in-human study with BYON4228, a humanized monoclonal antibody (mAb) directed against SIRPα.

DETAILED DESCRIPTION:
This study includes a dose escalation part (Part 1) in which the MTD and dose regimen for expansion (RDE) will be determined, and an expansion part (Part 2) to evaluate efficacy and safety in specific patient cohorts.

BYON4228 is a humanized IgG1 mAb directed against SIRPα. BYON4228 binds SIRPα expressed on innate immune cells, especially monocytes, macrophages and neutrophils. BYON4228 blocks binding of SIRPα to CD47 and inhibits signaling through the CD47-SIRPα axis.

ELIGIBILITY:
Inclusion Criteria:

* Part 1 (dose escalation): B-cell NHL expressing CD20 by immunohistochemistry (IHC) or flow cytometry, relapsed/refractory (R/R) to at least 2 prior lines of therapy.
* Part 2 (dose expansion):

A. Histologically confirmed diffuse large B-cell lymphoma (DLBCL) or Mantle Cell Lymphoma (MCL) expressing CD20 by IHC or flow cytometry, R/R to frontline therapy.

B. Histologically confirmed marginal zone or follicular lymphoma (Grade 1-3a) expressing CD20 by IHC or flow cytometry, R/R to at least 2 prior lines of therapy.

* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1;
* Adequate organ function;
* Laboratory measurements, blood counts (Growth Factor (GF) support and blood transfusions are not allowed within 2 weeks prior to this assessment):

  * Hemoglobin ≥ 8.5 g/dL (> 5.28 mmol/L);
  * Absolute neutrophil count (ANC) ≥ 1.0 × 10^9/mL;
  * Platelet counts ≥ 50 × 10^9/mL;

Exclusion Criteria:

* Having been treated with CD47 or SIRPα targeting agents at any time or other anticancer therapy within 4 weeks or as defined in the protocol;
* History of hypersensitivity or allergic reaction to any of the excipients of BYON4228 or rituximab which led to permanent discontinuation of the treatment;
* Burkitt's lymphoma;
* Red blood cell (RBC) transfusion dependence;
* Patients with active graft versus host disease (GVHD) or ongoing immunosuppression for GVHD;
* History of autoimmune hemolytic anemia or autoimmune thrombocytopenia;
* History of active autoimmune disorders (including but not limited to: Crohn's disease, rheumatoid arthritis, scleroderma, systemic lupus erythematosus, Grave's disease) or other conditions that compromise or impair the immune system (except for hypogammaglobulinemia);
* History (within 6 months prior to start IMP) or presence of clinically significant cardiovascular disease such as unstable angina, congestive heart failure, myocardial infarction, uncontrolled hypertension, or cardiac arrhythmia requiring medication;
* Currently diagnosed or suspected CNS involvement;
* Severe active infection or other severe uncontrolled systemic disease (e.g. advanced renal disease, pulmonary, uncontrolled diabetes mellitus, severely immunocompromised state, or metabolic disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2024-03-04 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities | 28 days
  Part 1

SECONDARY OUTCOMES:
Objective response rate | 2 years
  Part 2

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Koper, Study Director — Byondis B.V., The Netherlands
Locations (12):
- Italy (5):
  - ASST Spedali Civili di Brescia, Brescia
  - Istituto di Candiolo - Fondazione del Piemonte per l'Oncologia - IRCCS, Candiolo
  - Instituto Europeo di Oncologia, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRCCS IRST, Ravenna
- Netherlands (2):
  - Vrije Universiteit Medisch Centrum, Amsterdam
  - Radboud UMC, Nijmegen
- Spain (3):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Institut Català d'Oncologia, Barcelona
  - Centro Integral Oncológico Clara Campal (CIOCC) Hospital Universitario HM Sanchinarro, Madrid
- United Kingdom (2):
  - The Christie NHS Foundation Trust, Manchester
  - University Hospitals Plymouth NHS Trust, Plymouth

IPD SHARING:
Plan to Share IPD: No